CLINICAL TRIAL: NCT01312467
Title: A Phase IIa Trial of Metformin for Colorectal Cancer Risk Reduction Among Patients With a History of Colorectal Adenomas and Elevated Body Mass Index
Brief Title: Trial of Metformin for Colorectal Cancer Risk Reduction for History of Colorectal Adenomas and Elevated BMI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NCI-2011-01744; NCI-2011-01744 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); UCI 10-31 (Other: Chao Family Comprehensive Cancer Center); 2010-7705 (Other: UCIrvine); UCI09-13-01 (Other: DCP); P30CA062203 (NIH); N01CN35160 (NIH)
Record Dates: First submitted 2011-03-07; First posted 2011-03-10 (Estimated); Results first posted 2015-06-25 (Estimated); Last update posted 2019-03-05 (Actual); Status verified 2019-02

CONDITIONS: Adenomatous Polyp; Colorectal Cancer; Obesity
MeSH Terms: conditions — Adenomatous Polyps; Colorectal Neoplasms; Obesity | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Prevention (metformin hydrochloride) (Experimental): Patients receive metformin hydrochloride PO QD during week 1 and then BID during weeks 2-12. Treatment continues for 12 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: metformin hydrochloride

INTERVENTIONS:
Drug: metformin hydrochloride
  Other Names: Glucophage

SUMMARY:
The purpose of this study is to find out whether METFORMIN decreases protein markers in colorectal tissue. This is a phase IIA study of the pharmacodynamics, safety and tolerability of Metformin in decreasing colorectal mucosa in patients with a history of colorectal adenomas in the past 3 years and a BMI >= 30, with decimals rounded to the nearest whole integer. Metformin as a potential chemopreventive agent for inhibition of the relevant molecular pathways involved in human colorectal carcinogenesis.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if a 12-week intervention of oral metformin (metformin hydrochloride) treatment among obese patients with a history of colorectal adenomas results in at least a 35% decrease in colorectal mucosa activated pS6serine235 from baseline as assessed via immunostaining.

SECONDARY OBJECTIVES:

I. To assess the effect of metformin on additional relevant biomarkers in serum: metformin levels; fasting insulin-like growth factor (IGF)-1, insulin-like growth factor binding protein (IGFBP)-1, IGFBP-3; fasting leptin; fasting Adiponectin; fasting and 2 hour post-prandial insulin and glucose.

II. To examine the correlation among biomarkers (serum, tissue). III. To assess the independent effects of treatment on each biomarker, using multivariate regression models to account for clinical and biomarker data.

IV. To document the safety and tolerability of metformin in the study population.

TERTIARY OBJECTIVES:

I. To assess the effect of metformin on additional relevant biomarkers in tissue via immunostaining. This will include the effects on levels of colorectal mucosa proliferation estimated by: phosphorylated AMPK (pAMPK), phosphorylated AKTserine 473 (pAKT), phosphorylated mTOR, phosphorylated insulin receptor (pIR), phosphorylated IGF-1 (pIGF-1) receptor, and Ki-67.

II. To cross-validate immunostaining results with Western blotting experiments in a subset of consecutive patients for the following endpoints: phosphorylated S6serine235 (pS6serine235), phosphorylated AMPK (pAMPK), phosphorylated AKTserine 473 (pAKT), phosphorylated mTOR, phosphorylated insulin receptor (pIR), phosphorylated IGF-1 (pIGF-1) receptor, and Ki-67.

OUTLINE:

Patients receive metformin hydrochloride orally (PO) once daily (QD) during week 1 and then twice daily (BID) during weeks 2-12. Treatment continues for 12 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed up for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* History of prior colorectal adenomas within the past 3 years; only patients who have had adenomas endoscopically removed are eligible; documentation of colorectal adenomas must be determined via review of pathology reports
* Body mass index (BMI) >= 30; rounded to the nearest whole integer
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Leukocytes ≥ 3,000/μL (>= 2,500/μL for African-American participants)
* Absolute neutrophil count >= 1,500/μL (>= 1,000/μL for African-American participants)
* Platelets >= 100,000/μL
* Total bilirubin within normal institutional limits
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 1.5 X institutional upper limit of normal (ULN)
* Creatinine within normal institutional limits
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation
* A serum pregnancy test must be performed and be negative in all women of childbearing potential within 2 weeks prior to starting treatment
* Ability to understand and willingness to sign a written informed consent document

Exclusion Criteria:

* History of colorectal cancer or other cancer(s) (except for non-melanoma skin cancers) within the last 3 years
* Family history of hereditary intestinal polyp disorder (e.g., familial adenomatous polyposis [FAP], hereditary non-polyposis colorectal cancer [HNPCC], Putz-Jegher's disease)
* Participants with diabetes
* History of vitamin B12 deficiency or megaloblastic anemia
* History of lactic acidosis
* Diet or other medications for weight loss
* Diseases associated with weight loss: anorexia, bulimia, or nausea
* Treatment with medications that may increase metformin levels: cationic drugs, e.g., digoxin, amiloride, procainamide, trimethoprim, vancomycin, triamterene, and morphine
* Treatment with other oral hypoglycemic agents
* Participants who have undergone full bowel resection, ablation or other local therapies
* Participants may not be receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to metformin
* Participants with human immunodeficiency virus (HIV), cirrhosis of any cause, NASH (nonalcoholic steatohepatitis), or hepatitis (auto-immune or infectious)
* Kidney disease or renal insufficiency (defined as serum creatinine > 1.4 mg/dL for females or > 1.5 mg/dL for males)
* Metabolic acidosis, acute or chronic, including ketoacidosis
* Uncontrolled intercurrent illness including, but not limited to:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness/social situations that would limit compliance with study requirements
  * Renal failure
  * Hepatic failure
  * Sepsis
  * Hypoxia
* Pregnant or breastfeeding women are excluded
* Participants anticipating elective surgery during the study period
* Contraindication to colonoscopy/flexible sigmoidoscopy
* Participants may not be using metformin, cimetidine (Tagament) furosemide (Lasix), nifedipine (Cardizem), Ranitidine (Zinetac or Zantac), digoxin (Lanoxin), Quinidine or any other drug contraindicated for use with metformin
* Chronic alcohol use or a history of alcohol abuse
* Participants with any medical psychosocial condition that, in the opinion of the investigator, could jeopardize participation in and compliance with the study criteria
* Participants that regularly use aspirin (ASA), nonsteroidal anti-inflammatory drugs (NSAIDs), calcium, and cyclooxygenase (Cox)-2 inhibitors are not eligible for enrollment; however, patients that use aspirin 81 mg daily, or aspirin 325 mg, NSAIDs, calcium, or Cox-2 inhibitors at a frequency < 10 times per month are eligible

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2011-03; Primary Completion 2014-03 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Zell, Principal Investigator — University of California Medical Center At Irvine-Orange Campus
Locations (4):
- United States (3):
  - Veterans Administration Long Beach Medical Center, Long Beach, California
  - University of California Medical Center At Irvine-Orange Campus, Orange, California
  - Kaiser Permanente - Sacramento, Sacramento, California
- Jewish General Hospital, Montreal, Quebec, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between 2011 and 2013, 45 obese colorectal adenoma (CRA) patients were enrolled at three study sites: UC Irvine, Long Beach VAMC, and Kaiser Permanente, Sacramento).
Groups:
- Prevention (Metformin Hydrochloride): Patients receive metformin hydrochloride PO QD during week 1 and then BID during weeks 2-12. Treatment continues for 12 weeks in the absence of disease progression or unacceptable toxicity.
  metformin hydrochloride: Given PO
  pharmacological study: Correlative studies
  laboratory biomarker analysis: Correlative studies
Period: Overall Study
Arm/Group | Prevention (Metformin Hydrochloride)
Started | 45
Completed | 32
Not Completed | 13
Not completed — Adverse Event | 4
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 2
Not completed — Deported to country of origin | 1
Not completed — Another medical condition | 1
Not completed — Ineligible | 4

BASELINE CHARACTERISTICS:
Population: 45 participants were enrolled into the study
Arm/Group | Prevention (Metformin Hydrochloride)
Number analyzed (Participants) | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.6 (6.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 30
Region of Enrollment [Number; unit: participants]
  United States | 45

OUTCOME MEASURES:

1. Primary Outcome: Change in Activated S6serine235 (i.e., the Ratio of pS6serine235/S6serine235)
Description: Tissue S6Ser235 immunostaining was analyzed by the study pathologist using Histo Score (HScore) analysis at baseline and post- metformin (Week 12). The Hscore is determined by estimation of the percentage of cells positively stained with mild, moderate, or strong staining intensity. The final score is determined by weighted estimate, as follows: Hscore = (# cell stained with High intensity/total # cells)x3 + (# cells stained with median intensity/total # cells)x2 + (# cells stained with low intensity/total # cells)x1. Mean and standard deviation of the change in the histo score (H score) of pS6serine235 from baseline were calcuated.
Time Frame: From baseline to 12 weeks
Population: The analysis is based on 32 participants who have evaluable data.
Measure: Mean (Standard Deviation); unit: weighted ratio of staining cells
Arm/Group | Prevention (Metformin Hydrochloride)
Number analyzed (Participants) | 32
weighted ratio of staining cells | 0.0228 (0.444)
Statistical Analysis 1: Comparison: Prevention (Metformin Hydrochloride); Test type: Superiority or Other; p > 0.773, A paired t-test

2. Secondary Outcome: Effects of Metformin Hydrochloride on Colorectal Mucosa Proliferation (Ki-67, Phosphorylated IGF-1 Receptor, Phosphorylated Insulin Receptor, Phosphorylated AKT, Phosphorylated mTOR, and Phosphorylated AMP Kinase)
Description: Data not collected.
Time Frame: Up to 16 weeks
Population: Funding was not secured to complete the secondary and tertiary endpoints.
Groups:
- Prevention (Metformin Hydrochloride): Patients receive metformin hydrochloride PO QD during week 1 and then BID during weeks 2-12. Treatment continues for 12 weeks in the absence of disease progression or unacceptable toxicity.
  metformin hydrochloride
Arm/Group | Prevention (Metformin Hydrochloride)
Number analyzed (Participants) | 0

3. Secondary Outcome: Effects of Metformin Hydrochloride on Serum (Fasting and 2 Hour Postprandial Insulin and Glucose, Fasting IGF-1, IGFBP-1, IGFBP-3, Leptin, Adiponectin and Metformin Levels)
Description: Data not collected.
Time Frame: Up to 16 weeks
Population: Funding was not secured to complete the secondary and tertiary endpoints.
Arm/Group | Prevention (Metformin Hydrochloride)
Number analyzed (Participants) | 0

4. Secondary Outcome: Safety and Tolerability of Metformin Hydrochloride Treatment
Description: All participants will be evaluable for toxicity from the time of their first dose of metformin. Since toxicities in this study are measured as categorical data, primary analysis shall be by tests of binomial proportions (e.g., Mantel-Haenszel chi-squared statistic). This study will utilize the CTCAE (NCI Common Terminology Criteria for Adverse Events) Version 4.0 for toxicity and Serious Adverse Event reporting.
Time Frame: Up to 16 weeks
Population: 45 participants were enrolled and 45 participants were analyzed for toxicity.
Measure: Number; unit: adverse events
Arm/Group | Prevention (Metformin Hydrochloride)
Number analyzed (Participants) | 45
adverse events
  Grade 1 | 186
  Grade 2 | 23
  Grade 3 or higher | 1

ADVERSE EVENTS:
Time Frame: Adverse Events that were occurred on and after the treatment began date to the end of the study (up to 16 weeks).
Arm/Group | Prevention (Metformin Hydrochloride)
Serious Adverse Events (participants affected / at risk) | 1/45
Other Adverse Events (participants affected / at risk) | 36/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prevention (Metformin Hydrochloride) (N=45)
DUCTAL CARCINOMA IN SITU, HIGH GRADE, SOLID AND CRIBRIFORM TYPE WITH APOCRINE FEATURES AND FOCAL NEC (Reproductive system and breast disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prevention (Metformin Hydrochloride) (N=45)
ABDOMINAL CRAMPING (Gastrointestinal disorders) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
BLOATING (Gastrointestinal disorders) | 1 (1)
COLD (Infections and infestations) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 5 (5)
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1)
CRAMPING (Gastrointestinal disorders) | 3 (8)
CRAMPS IN LEGS (Musculoskeletal and connective tissue disorders) | 1 (2)
DECREASED HEARING (Ear and labyrinth disorders) | 1 (1)
DIARRHEA (Gastrointestinal disorders) | 14 (25)
DIFFICULTY HOLDING BLADDER-URGENCY (Renal and urinary disorders) | 1 (1)
DIZZINESS (Nervous system disorders) | 7 (7)
DRY MOUTH (Gastrointestinal disorders) | 3 (3)
DRY SKIN (Skin and subcutaneous tissue disorders) | 1 (1)
ELEVATED TEMPERATURE (General disorders) | 1 (2)
EYE IRRITATION (Eye disorders) | 1 (1)
FATIGUE (General disorders) | 7 (7)
FEELS AWAKE (Psychiatric disorders) | 1 (1)
FELT COLD (General disorders) | 1 (1)
FEVER (General disorders) | 2 (3)
FLATULENCE (Gastrointestinal disorders) | 8 (8)
HEADACHE (Nervous system disorders) | 5 (5)
HEARTBURN (Gastrointestinal disorders) | 5 (6)
HEAT RASH (Skin and subcutaneous tissue disorders) | 1 (1)
HEEL PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
HEMATOCHEZIA (Gastrointestinal disorders) | 1 (1)
HEMATOCRIT LAB RESULT BELOW THE NORMAL RANGE (Blood and lymphatic system disorders) | 1 (4)
HEMOGLOBIN LAB RESULT BELOW THE NORMAL RANGE (Blood and lymphatic system disorders) | 1 (4)
HEMORRHOIDS (Gastrointestinal disorders) | 1 (1)
HYPERTENSION (Vascular disorders) | 1 (1)
HYPOGLYCEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPOGLYCEMIC (Metabolism and nutrition disorders) | 1 (1)
INCREASED APPETITE (Metabolism and nutrition disorders) | 1 (1)
INCREASED GAS (Gastrointestinal disorders) | 1 (1)
INCREASED SWEATING (Skin and subcutaneous tissue disorders) | 1 (1)
INFECTION IN SITE OF LUMPECTOMY (Infections and infestations) | 1 (1)
INSOMNIA (Psychiatric disorders) | 3 (3)
IRON LAB RESULT OUT OF RANGE (Blood and lymphatic system disorders) | 1 (1)
ITCHY SKIN (Skin and subcutaneous tissue disorders) | 1 (1)
ITCHY THROAT (Respiratory, thoracic and mediastinal disorders) | 1 (2)
JITTERS (Nervous system disorders) | 1 (2)
KNEE PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
LEG CRAMPS (Musculoskeletal and connective tissue disorders) | 2 (2)
LIGHTHEADED (Nervous system disorders) | 2 (2)
LIGHTHEADED/DIZZINESS (Nervous system disorders) | 1 (2)
LIGHTHEADEDNESS (Nervous system disorders) | 2 (2)
LOOSE STOOLS (Gastrointestinal disorders) | 4 (4)
LOOSE STOOLS/DIARRHEA (Gastrointestinal disorders) | 1 (1)
LOSS OF APPETITE (Metabolism and nutrition disorders) | 6 (6)
LOSS OF APPETITE-EATING LESS (Metabolism and nutrition disorders) | 1 (1)
MILD CRAMPING (Gastrointestinal disorders) | 2 (5)
MILD GERD (Gastrointestinal disorders) | 1 (1)
MORE BRUISING (Injury, poisoning and procedural complications) | 1 (1)
MUSCLE PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
NASAL CONGESTION (Infections and infestations) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 7 (8)
SCIATICA FLARE (Musculoskeletal and connective tissue disorders) | 1 (1)
SCRATCHED LEFT EYE CORNEA (Eye disorders) | 1 (1)
SHORTNESS OF BREATH (Respiratory, thoracic and mediastinal disorders) | 2 (2)
SLIGHT COLD (General disorders) | 1 (1)
SMALLER APPETITE (Metabolism and nutrition disorders) | 1 (1)
SORE RIGHT WRIST (Musculoskeletal and connective tissue disorders) | 1 (1)
STOMACH CRAMPS (Gastrointestinal disorders) | 1 (1)
STOMACH DISCOMFORT (Gastrointestinal disorders) | 1 (1)
STOMACH PAIN (Gastrointestinal disorders) | 6 (7)
STUFFY NOSE (Respiratory, thoracic and mediastinal disorders) | 1 (1)
SWEATING (Skin and subcutaneous tissue disorders) | 2 (2)
SWEET CRAVINGS (Metabolism and nutrition disorders) | 1 (1)
SWELLING LESS IN FEET (General disorders) | 1 (1)
TRANSFERRIN SATURATION OUT OF RANGE - LOW (Blood and lymphatic system disorders) | 1 (1)
TWITCHING RIGHT THIGH (Musculoskeletal and connective tissue disorders) | 1 (1)
VERY LOOSE STOOLS (Gastrointestinal disorders) | 1 (1)
VOMITING (Gastrointestinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less